CLINICAL TRIAL: NCT06484738
Title: Spatially Resolved IBD: Spatial Transcriptomics of Inflammatory Bowel Disease (IBD)
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: BGI, China (Other)
Responsible Party: Principal Investigator, Silvio Danese, Professore, IRCCS San Raffaele
Other Study IDs: STOmics
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Patients With Histologically Confirmed CD Undergoing Intestinal Resection According to Standard of Care Due to Complicating Disease; Patients With Histologically Confirmed UC Undergoing Intestinal Resection According to Standard of Care Due to Complicating Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with histologically confirmed CD: patients with histologically confirmed CD undergoing intestinal resection
  Interventions: Other: transcriptomic analysis
- patients with histologically confirmed UC: patients with histologically confirmed UC undergoing intestinal resection
  Interventions: Other: transcriptomic analysis

INTERVENTIONS:
Other: transcriptomic analysis — to use their biological samples from UC and CD patients, already stored at -80°C for transcriptomic analysis through STOmics Stereoseq

SUMMARY:
The goal of this retrospective observational study is to obtain the spatial resolution of the entire intestinal fibrotic process through the technology STOmics Stereoseq. For this study we will use surgical specimens from 8 UC e 8 CD previously collected for the already approved project, IBD Biobank, and stored at -80° C.

DETAILED DESCRIPTION:
This is a monocentric observational study in which we will use the biological material from surgery carried out for normal clinical practice, and already stored at -80°C.

This project has as purpose:

1. To unravel the changes in the intestine leading to complications in CD and UC patients. In particular, we aim to identify the cell populations, their spatial organization, interactions, and specific transcriptional shifts, leading the progression from healthy tissue to inflamed and from inflamed to fibrotic tissue. We will be interested in producing a profile of Spatial transcriptomics of all areas of the surgical specimen.
2. To compare the spatial organization and differential gene expression of tissue

ELIGIBILITY:
Inclusion Criteria:

* adult patient (age ≥18 years), both male and female patients with histologically confirmed CD and UC undergoing intestinal resection according to standard of care due to complicating disease, regardless of their current or past medical treatment;
* patients that have signed the IBD Biobank informed consent and consented to the use of their own biological material in future study or pertaining to the same field of investigation.

Exclusion Criteria:

* - patients with unconfirmed both UC and CD diagnoses;
* patients with superimposed dysplasia or cancer diagnosis and resections for which post- operative endoscopic assessment of recurrence is not feasible;
* patients who have not signed the IBD Biobank informed consent.

Ages: 18 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective observational study involving patients with Crohn's disease (CD) (n=8) and patients with ulcerative colitis (UC)(n=8) who had undergone surgery according to the standard of care. We will use the biological material from surgery carried out for normal clinical practice, and already stored at -80°C for IBD Biobank project. The retrospective referral period of time goes from July 2022 until July 2023.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Profile of Spatial transcriptomics of all areas of the surgical specimen from UC and CD patients | 1 year
  to perform a transcriptomic analysis of the entire surgical specimen will be embedded in OCT block. To overcome any failures in the OCT embedding, we will cut serial sections and stain them to evaluate the presence of all intestinal regions of interest, and then choose the adjacent one for the spatial analysis. Moreover, we will evaluate by histological assessment whether one single piece of surgical specimen will encompass not inflamed, inflamed (in case of UC) and also fibrotic areas (in case of CD)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan
  - Irccs Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No